CLINICAL TRIAL: NCT03217461
Title: A Non-randomized Controlled Clinical Trial of Corneal Autograft for Limbal Dermoid
Brief Title: Corneal Autograft for Limbal Dermoid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chunxiao Wang (Other)
Responsible Party: Sponsor-Investigator, Chunxiao Wang, Clinical investigator, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020KYPJ206
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Corneal Dermoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Limbal autograft (Experimental): Corneal dermoid tumor resection combined with femtosecond laser assisted limbal autograft
  Interventions: Procedure: Limbal autograft; Device: Femtosecond laser

INTERVENTIONS:
Procedure: Limbal autograft — Simple dermoid excision will be performed, followed by closure of the bare sclera and cornea by sutured femtosecond laser-assisted limbal autograft.
Device: Femtosecond laser — A commercial femtosecond laser to create a particular shaped graft for transplantation

SUMMARY:
To investigate the clinical efficacy of femtosecond laser-assisted autologous lamellar keratoplasty in treating corneal dermoids.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 5 to 35 years old,
2. Patients with limbal dermoid, scheduled for elective surgical excision,
3. The distance of less than 5 mm of lesion encroachment into the cornea,
4. The participant or their legal guardian has voluntarily chosen to participate in this study, has signed the informed consent form, and has demonstrated a high level of adherence to the study protocols and cooperation throughout the follow-up process.

Exclusion Criteria:

1. Keratoconus,
2. High myopia with a spherical equivalent of -15.0 D or less,
3. Ocular and facial active inflammation such as keratitis, trachoma, dacryocystitis, blepharitis, meibomian gland dysfunction, Sjogren's syndrome, cicatricial pemphigoid etc,
4. Corneal or ocular surface infection within 30 days prior to study entry,
5. Severe cicatricial eye disease,
6. Ocular surface malignancy,
7. Ocular comorbidities that affect the prognosis of transplantation, such as advanced glaucoma or retinal diseases,
8. History of allo-limbal transplantation, penetrating keratoplasty or anti-glaucoma filtering surgeries,
9. Uncontrolled diabetes with most recent Hemoglobin A1c greater than 8.5%,
10. Renal failure with creatinine clearance< 25ml/min,
11. Alanine aminotransferase > 40IU/L, or aspartate aminotransferase > 40IU/L,
12. Platelet levels < 150,000 or > 450,000 per microlite,
13. Hemoglobin < 12.0 g/dL (male) or < 11.0 g/dL (female),
14. Prothrombin time > 16s and activated partial thrombin time > 35s in patients not accepting anticoagulant therapy, An international normalized ratio greater than 3 in patients accepting anticoagulant therapy,
15. Pregnancy (positive test) or lactation,
16. Active immunological diseases,
17. Signs of current infection, including fever and treatment with antibiotics,
18. Participation in another simultaneous medical investigation or clinical trial.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Corneal Thickness | 1 week, 1 month, 3 months, 6 months, 9 months, 12 months and 18 months postoperatively
  To measure corneal thickness using anterior segment optical coherence tomography.
Corneal Transparency | Preoperatively, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months and 18 months postoperatively
  The transparency and appearance of the cornea will be observed using slit-lamp microscopy

SECONDARY OUTCOMES:
Best corrected visual acuity | Preoperatively, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months and 18 months postoperatively
  To measure best corrected visual acuity using ETDRS chart or Teller Acuity Cards.
Corneal power, astigmatism and aberration | Preoperatively, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months and 18 months postoperatively
  To measure the changes of corneal power, astigmatism and aberration using autorefractor keratometer and wavefront aberrometer respectively.
Cosmetic improvement | Preoperatively, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months and 18 months postoperatively
  A grading system from 0 to 4 with slit-lamp photographs will be used to determine cosmetic result of each graft.

OTHER OUTCOMES:
Restoration of corneal surface | 1 week, 1 month, 3 months, 6 months, 9 months, 12 months and 18 months postoperatively
  Restoration of a completely epithelized, stable, and avascular corneal surface.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Ting Huang, M.D.Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No